CLINICAL TRIAL: NCT06191666
Title: Design and Integration of a Survivorship Nutrition Intervention Into an Established Exercise Oncology Program: the BfedBwell Pilot Intervention
Brief Title: BfedBwell Proof-of-Concept Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1501.cc
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cancer Survivorship; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer Survivors (Experimental): Cancer survivors with ow/ob who have completed active treatment will take part in a single-arm 12-week feasibility/acceptability/proof-of-concept study incorporating group nutrition education and discussion, skills development sessions and cooking demonstrations, and 1:1 counseling with a dietitian.
  Interventions: Behavioral: Group-based education and discussion; Behavioral: Individual 1:1 counseling; Behavioral: Group based behavioral skills development and cooking demonstrations; Behavioral: BfitBwell

INTERVENTIONS:
Behavioral: Group-based education and discussion — Group-based education and discussion (60 minutes each per week, virtual and in-person) based upon guidelines for nutrition for cancer survivorship (e.g., follow a plant-based diet with a variety of vegetables, fruits, whole grains, and legumes; limit alcohol intake; reduce consumption of highly processed foods and foods high in salt; achieve a weekly calorie deficit of approximately 3500 kcal for weight loss)
Behavioral: Individual 1:1 counseling — Individual 1:1 counseling sessions (30 minutes each per month, virtual) with an RD to review progress and address barriers
Behavioral: Group based behavioral skills development and cooking demonstrations — Group-based behavioral skills development sessions and cooking demonstrations (60-90 minutes each per month, in-person) to focus on behavior change techniques (e.g., self-monitoring, goal setting) and nutrition skills (e.g., recipe development, label reading).
Behavioral: BfitBwell — This program consists of a supervised exercise program developed by a cancer exercise specialist and based upon the NCCN guidelines for physical activity during cancer survivorship and other recommendations.

SUMMARY:
This single-arm proof-of-concept pilot will assess the feasibility and acceptability of integrating a survivorship nutrition intervention (BfedBwell) into an existing clinical exercise oncology program (BfitBwell).

DETAILED DESCRIPTION:
Individuals with experience in delivery of lifestyle (e.g., diet, physical activity) interventions will be recruited to deliver and evaluate the integrated BfedBwell + BfitBwell intervention.

Cancer survivors with overweight/obesity who have completed active treatment will be recruited from the University of Colorado Anschutz Medical Campus for participation in a 12-week single-arm study of the integrated BfedBwell + BfitBwell intervention. Feasibility and acceptability will be evaluated. Exploration of intervention effect on adherence to cancer survivorship guidelines, body composition, and cardiometabolic indicators of health will be used to evaluate proof-of-concept prior to advancing to efficacy testing.

ELIGIBILITY:
Inclusion Criteria:

For program delivery staff:

1. Men and women
2. Age ≥ 18 years
3. Speak English
4. Self-reported previous experience in the delivery of nutrition, exercise, or behavioral weight management programs

For intervention participants:

1. Men and women
2. Age 18-75 years
3. Body Mass Index 25-45 kg/m2
4. Completion of active cancer therapy with curative intent at least three months and no more than five years prior to enrollment; ongoing hormone therapy is permitted
5. Have a primary care provider (or are willing to establish care with a primary care provider prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions and who will provide clearance to participate in a nutrition and exercise program
6. Ability and willingness to participate in a supervised exercise program; with ability assessed by the Physical Activity Readiness Questionnaire (PAR-Q+) and questions based upon National Comprehensive Cancer Network guidelines (note: any positive responses will trigger a required physician clearance form)
7. Speak English
8. Have access to a computer or smart phone and Internet
9. Live or work within 30 miles of the Anschutz Health and Wellness Center (exceptions may be made at the discretion of the study PI on a case-by-case basis for highly motivated subjects)
10. Not be planning to travel for >2 consecutive weeks or relocate/move during the intervention
11. Agree to refrain from use of all nutritional supplements aside from those prescribed by a physician for the duration of the study
12. Capable and willing to give informed consent and understand exclusion criteria
13. Willing to attend weekly small group sessions (behavioral skills development and/or group support) and/or 1:1 counseling held by a registered dietitian (RD) and attend up to two BfitBwell exercise sessions per week
14. Not meeting dietary guidelines [i.e., Healthy Eating Index (HEI) score <80 as assessed via National Cancer Institute Diet History Questionnaire III (NCI DHQ III) food frequency questionnaire] or physical activity guidelines [i.e., <150 minutes moderate/vigorous activity per week via self-report on Godin-Shephard Leisure-Time Physical Activity Questionnaire]

Exclusion Criteria:

For program delivery staff:

None

For intervention participants:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status 2 or higher
2. Actively undergoing cancer therapy or within 3 months of completion of surgery, chemotherapy, or radiation treatment
3. Greater than 5 years post-active therapy
4. Plans to relocate within the next 6 months
5. Plans for extended travel (>2 weeks) within the next 6 months
6. For females:

   1. Currently pregnant or lactating
   2. Pregnant within the past 6 months
   3. Planning to become pregnant in the next 18 months; sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception
7. Any major surgery within the past 3 months, including mastectomy
8. Have completed treatment that significantly impacts digestion, metabolism, and/or food intake (e.g., surgical loss of esophagus, stomach, colon)
9. Recent (past 6 months) acute coronary event, unstable angina, coronary revascularization, stroke, or pulmonary embolism
10. Symptoms suggestive of cardiovascular disease (e.g., chest pain, shortness of breath at rest or with mild exertion, lightheadedness, syncope)
11. Uncontrolled hypertension, defined as diastolic blood pressure >100 mmHg, systolic blood pressure >160 mmHg, or resting heart rate >100 bpm as measured in duplicate on the screening visit after 5 minutes of rest in a seated position (if screening is needed due to lack of updated medical record within previous 12 months)
12. Diabetes (history of type 1 or type 2 diabetes, hemoglobin A1c >7.5%, or fasting glucose ≥126 mg/dL as measured during the screening visit if screening is needed due to lack of updated medical record within previous 12 months) unless well controlled on metformin alone
13. History of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen is acceptable
14. Triglycerides >500 mg/dL as measured on the screening visit (if screening is needed due to lack of updated medical record within previous 12 months)
15. LDL cholesterol >200 mg/dL as measured on the screening visit (if screening is needed due to lack of updated medical record within previous 12 months)
16. Presence or history of other metabolic or chronic health problems which would impact ability to safely participate in a weight loss intervention involving diet and exercise: significant cardiac arrhythmias or cardiac valvular disease, significant gastrointestinal, pulmonary, renal, musculoskeletal, neurologic, hematologic, or psychiatric disease
17. Have started lipid-lowering, hypertension, or oral hypoglycemic medication in previous 3 months
18. Sustained use of prescription or over-the-counter medications known to significantly impact appetite, weight, or energy metabolism (e.g., obesity pharmacotherapeutics agents, appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants) with the exception of anti-endocrine or Her2 directed treatment for breast cancer and standard of care anti-emetic or anti-diarrheal agents.
19. Sustained use of systemic glucocorticoids (current or in the past 6 months) unless physiologic replacement therapy for adrenal insufficiency
20. Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed >1 year before screening, (2) lap banding if the band has been removed >1 year before screening, (3) intragastric balloon if the balloon has been removed >1 year before screening, (4) duodenal-jejunal bypass sleeve if the sleeve has been removed >1 year before screening, or (5) AspireAssist or other endoscopically placed weight loss device if the device has been removed >1 year before screening
21. Participation within previous 6 months, current participation in, or planning to participate in any formal nutrition, weight loss, or physical activity programs or clinical trials over the next 6 months
22. Previous participation the BfitBwell exercise oncology program
23. Current alcohol or substance abuse as assessed by the Cut down, Annoyed, Guilty, and Eye-Opener (CAGE) questionnaire (note: study PI will follow up if screener raises any concerns of substance abuse to determine final eligibility)
24. History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS-26) or pattern of response on the Questionnaire of Eating and Weight Patterns (QEWP-5) suggestive of possible binge eating disorder or bulimia will require further assessment by the study MD to determine if it is appropriate for the subject to participate in the study
25. Current severe depression or history of severe depression within the previous year, based on Center for Epidemiologic Studies Depression Scale (CES-D)
26. History of other significant psychiatric illness (e.g., psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the study MD would interfere with ability to adhere to the diet and exercise interventions
27. Have medical or physical limitations or contraindications to engaging in physical activity (e.g., severe orthopedic conditions, paralysis) or are considered high-risk based on American College of Sports Medicine (ACSM) guidelines
28. Are cognitively unable to consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Determine the research protocol recruitment feasibility of the BfedBwell nutrition intervention | 12 weeks
  Recruitment will be assessed as the number of adults screened and the proportion of eligible screens who enroll.
Determine the research protocol adherence feasibility of the BfedBwell nutrition intervention | 12 weeks
  Adherence will be assessed as [# sessions attended/# sessions provided]
Determine the research protocol outcome assessment feasibility of the BfedBwell nutrition intervention | 12 weeks
  Outcome assessment rates will be assessed as [# completing assessments/# enrolled].
Determine the research protocol retention feasibility of the BfedBwell nutrition intervention | 12 weeks
  Retention will be assessed as [# of participants who complete the 12-week intervention/# of participants enrolled].
Determine the intervention feasibility by program delivery staff using Feasibility of Intervention Measure (FIM) | 12 weeks
  Upon completion of the intervention, program delivery staff will be asked to complete the Feasibility of Intervention Measure (FIM). A Likert scale from 1 (completely disagree) to 5 (completely agree) is used for each question; higher scores indicate greater intervention feasibility.
Determine the intervention acceptability by program delivery staff using Acceptability of Intervention Measure (AIM) | 12 weeks
  Upon completion of the intervention, program delivery staff will be asked to complete the Acceptability of Intervention Measure (AIM). A Likert scale from 1 (completely disagree) to 5 (completely agree) is used for each question; higher scores indicate greater intervention acceptability.
Determine the intervention acceptability by program delivery staff using Intervention Appropriateness Measure (IAM) | 12 weeks
  Upon completion of the intervention, program delivery staff will be asked to complete the Intervention Appropriateness Measure (IAM). A Likert scale from 1 (completely disagree) to 5 (completely agree) is used for each question; higher scores indicate greater intervention appropriateness.
Determine the intervention acceptability by participants using the Net Promoter Score (NPS) | 12 weeks
  Participants will be asked to complete weekly ratings using the Net Promoter Score (NPS). Respondents are grouped as follows: 1) promoters (score 9-10) are loyal enthusiasts who will keep referring others and fueling growth, 2) passives (score 7-8) are satisfied but unenthusiastic customers who are vulnerable to competitive offerings, and 3) detractors (score 0-6) are unhappy customers who can impede growth with negative word-of-mouth. The final NPS score is calculated as % promoters - % detractors. NPS scores range from -100 to +100, with scores >0 indicating good acceptability.
Determine the intervention acceptability by participants and program providers during qualitative interviews | 12 weeks
  1:1 interviews will be conducted with all program delivery staff and BfedBwell survivorship nutrition intervention participants after the 12-week intervention to assess acceptability of intervention and provide feedback for continued refinement.

SECONDARY OUTCOMES:
Assess preliminary efficacy for increased adherence to lifestyle recommendations | 12 weeks
  Determine the change in adherence to cancer survivorship guidelines as measured by World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) scoring criteria. Scores range from 0 to 7 points. A higher score reflects greater adherence to the recommendations.
Assess preliminary efficacy for weight loss | 12 weeks
  Determine the change in weight as measured by digital scale. A lower weight indicates an improvement.
Assess preliminary efficacy for improvement in body composition | 12 weeks
  Determine the change in body composition as measured by dual x-ray absorptiometry (DXA). A lower body fat percentage indicates an improvement.
Measure the change in systolic blood pressure to determine improved cardiometabolic health | 12 weeks
  Systolic blood pressure will be measured at specific time points during the trial. A lower systolic blood pressure indicates an improvement.
Measure the change in diastolic blood pressure to determine improved cardiometabolic health | 12 weeks
  Diastolic blood pressure will be measured at specific time points during the trial. A lower diastolic blood pressure indicates an improvement.
Measure changes in total cholesterol to determine improved cardiometabolic health | 12 weeks
  Total cholesterol will be measured at specific time points during the trial. A lower total cholesterol indicates an improvement.
Measure changes in LDL cholesterol to determine improved cardiometabolic health | 12 weeks
  LDL cholesterol will be measured at specific time points during the trial. A lower LDL cholesterol indicates an improvement.
Measure changes in HDL cholesterol to determine improved cardiometabolic health | 12 weeks
  HDL cholesterol will be measured at specific time points during the trial. A higher HDL cholesterol indicates an improvement.
Measure changes in triglycerides to determine improved cardiometabolic health | 12 weeks
  Triglycerides will be measured at specific time points during the trial. Lower triglycerides indicate an improvement.
Measure changes in glucose to determine improved cardiometabolic health | 12 weeks
  Glucose levels will be measured at specific time points during the trial. Lower glucose levels indicate an improvement.
Measure changes in insulin to determine improved cardiometabolic health | 12 weeks
  Insulin levels will be measured at specific time points during the trial. Lower insulin levels indicate an improvement.
Intervention safety determined by number of adverse events | 12 weeks
  Overall rates of study-related mild, moderate, severe, and serious adverse events (AEs) will be tracked by study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Emily B Hill, PhD, RDN, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States